CLINICAL TRIAL: NCT04209426
Title: Etude de Cohorte Observationnelle Rétrospective SYMBOL CUP 2
Brief Title: Retrospective Observational Cohort Study of SYMBOL CUP DM 2
Acronym: SYMCOR-2
Status: Completed | Type: Observational
Sponsor: Dedienne Sante S.A.S. (Industry)
Responsible Party: Sponsor
Other Study IDs: SYMCOR-2
Record Dates: First submitted 2019-12-20; First posted 2019-12-24 (Actual); Results first posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-02

CONDITIONS: Revision Total Hip Arthroplasty; Primary Total Hip Arthroplasty
Keywords: total hip arthroplasty; complex; revision; hemispherical dual-mobility acetabular cup; safety; efficacy; implant survival; prosthetic dislocation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HMB-DMR-HA: Total hip arthroplasty with hemispherical metal-back dual-mobility acetabular cup with tripod fixation consisting of a hydroxyapatite-coated outer surface as well as two pegs and one screw.
  Interventions: Device: THA with SYMBOL CUP DMR HA
- HMB-DM-CEM: Total hip arthroplasty with hemispherical metal-back dual-mobility acetabular cup with tripod fixation consisting of a bare metal outer surface to be covered with bone-compatible cement.
  Interventions: Device: THA with SYMBOL CUP DM CEM

INTERVENTIONS:
Device: THA with SYMBOL CUP DMR HA
  Groups: HMB-DMR-HA
Device: THA with SYMBOL CUP DM CEM
  Groups: HMB-DM-CEM

SUMMARY:
This is a single-center retrospective observational cohort study of consecutively operated patients who underwent total hip arthroplasty (THA) with a SYMBOL CUP DMR HA or a SYMBOL CUP DM CEM hemispherical dual mobility acetabular implant. The purpose of this study is to estimate the safety and efficacy of those two implants at two-year follow-up.

DETAILED DESCRIPTION:
Description according to PICOS (Patient, Intervention, Comparator, Outcomes, Study design) framework:

Patients:

- Adult men and women requiring a total hip arthroplasty

Intervention:

- THA with SYMBOL CUP DMR HA or SYMBOL CUP DM CEM hemispherical dual mobility acetabular implants.

Comparator: None

Outcomes:

* Safety 1: Implant survival over 2-year follow-up.
* Safety 2: All adverse events, with focus on implant dislocation, infections, revision surgery
* Efficacy 1: Harris Hip Score (HHS) at baseline and 1-year follow-up.
* Efficacy 2: Modified HHS (mHHS) consisting of pain + functional subscores at baseline, 1-year and 2-year follow-ups.
* Efficacy 2: Devane score at baseline, 1-year and 2-year follow-ups.
* Efficacy 3: Charnley classification at baseline, 1-year and 2-year followups.

Study design:

* single-center retrospective observational cohort study of consecutively operated patients who underwent total hip arthroplasty 2 years prior to study start.
* Prospective 2-year follow-up letter and phone questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* All patients with total hip implant using hemispheric dual-mobility SYMBOL CUP DMR HA or SYMBOL CUP DM CEM
* Operation performed by the primary investigator
* Delay between index operation and March 1 2018 has reached 2 years

Exclusion Criteria:

* patient refusal to participate in the study
* minors (age < 18 years)
* patients under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Exhaustive recruitment of patients meeting inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-03-18 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Estour, M.D., Principal Investigator — Hôpital Privé Medipole de Savoie
Locations (1):
- Hôpital Privé Medipole de Savoie, Challes-les-Eaux, France

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- HMB-DMR-HA: Total hip arthroplasty with hemispherical metal-back dual-mobility acetabular cup with tripod fixation consisting of a hydroxyapatite-coated outer surface as well as two pegs and one screw.
  THA with SYMBOL CUP DMR HA
- HMB-DM-CEM: Total hip arthroplasty with hemispherical metal-back dual-mobility acetabular cup with tripod fixation consisting of a bare metal outer surface to be covered with bone-compatible cement.
  THA with SYMBOL CUP DM CEM
Period: Overall Study
Arm/Group | HMB-DMR-HA | HMB-DM-CEM
Started | 15 | 5
Completed | 12 | 3
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HMB-DMR-HA | HMB-DM-CEM | Total
Number analyzed (Participants) | 15 | 5 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.3 (33.4) | 77.6 (6.7) | 77.4 (26.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 12
  Male | 6 | 2 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 15 | 5 | 20
BMI [Mean (Standard Deviation); unit: Kg/m2] | 24.4 (4.8) | 25.8 (2.4) | 24.8 (4.2)
Operated side [Count of Participants; unit: Participants]
  Right | 10 | 2 | 12
  Left | 5 | 3 | 8
Type of surgery [Count of Participants; unit: Participants]
  THA | 5 | 0 | 5
  rTHA | 10 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Implant Survival: Acetabular Cup Survival at 2-year Follow-up
Description: This is a the ratio of the number of patient joints surviving with the acetabular prosthesis in position at a given follow-up time (numerator) over the initial number of those joints from the date they received the acetabular prosthesis (denominator). The cumulative ratio is recalculated at each event using the Kaplan-Meier method from the date of each joint index operation through the date of each participant's death or prosthetic removal surgery or loss-to-follow-up or last assessment alive with the acetabular prosthesis in place. The longest duration between the index operation and the final assessment is 2 years.
Time Frame: 2 years as of index operation
Measure: Number (95% Confidence Interval); unit: percentage of implants survival
Arm/Group | HMB-DMR-HA | HMB-DM-CEM
Number analyzed (Participants) | 15 | 5
percentage of implants survival | 94.7 [68.1 to 99.2] | 100 [100 to 100]

2. Secondary Outcome: Number of Patients With One or Several Post-operative Adverse Events and Count of Each Serious Adverse Event and Aggregate Count of Adverse Events
Description: All serious post-operative adverse events are taken into account including implant dislocation, infections, revision surgery.
Time Frame: 2 years as of index operation
Measure: Number; unit: participants
Arm/Group | HMB-DMR-HA | HMB-DM-CEM
Number analyzed (Participants) | 15 | 5
participants | 10 | 0

3. Secondary Outcome: Harris Hip Score (HHS) at Baseline and 1-year Follow-up
Description: Harris Hip Score (HHS) is measured at each assessment in each patient. HHS is a physician-completed instrument that consists of subscales for pain severity (1 item, 0-44 points), function (7 items, 0-47 points), absence of deformity (1 item, 0-4 points), and range of motion (2 items, 0-5 points). Scores range from 0 (worse disability) to 100 (less disability).
  The mean and confidence interval of the score is measured at each assessment as well as for the within-patient difference between assessments
Time Frame: 1 year as of index operation
Population: Number at stake at 1 year take into account the following events (death, lost to follow-up and revisions)
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | HMB-DMR-HA | HMB-DM-CEM
Number analyzed (Participants) | 15 | 5
score on a scale
  HHS preoperative | 34 (37.7) | 58 (13.8)
  HHS 1-year: number analyzed (Participants) | 11 | 5
  HHS 1-year | 89 (24) | 86 (34.2)

4. Secondary Outcome: The Modified Harris Hip Score (Modified HHS) at Baseline, 1-year and 2-year Follow-up
Description: The modified Harris Hip Score (modified HHS) is the sum of pain subscore and functional subscore of the Harris Hip Score. It consists of subscales for pain severity (1 item, 0-44 points), function (7 items, 0-47 points). Scores range from 0 (worse disability) to 91 (less disability)The score is measured at each assessment in each patient. The mean and confidence interval of the score is measured at each assessment as well as for the within-patient difference between assessments
Time Frame: 2 years as of index operation
Population: Number at stake at 1 year or 2-years take into account the following events (death, lost to follow-up and revisions)
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | HMB-DMR-HA | HMB-DM-CEM
Number analyzed (Participants) | 15 | 5
score on a scale
  mHHS preoperative | 29 (21.5) | 49 (13.4)
  mHHS 1-year: number analyzed (Participants) | 11 | 5
  mHHS 1-year | 80 (22.5) | 77 (34.2)
  mHHS 2-year: number analyzed (Participants) | 9 | 3
  mHHS 2-year | 87 (11.3) | 80 (10.0)

ADVERSE EVENTS:
Time Frame: Collection of all side-effects occurring between surgery (prosthesis insertion) and the last clinical follow-up (2-year follow-up at least)
Arm/Group | HMB-DMR-HA | HMB-DM-CEM
All-Cause Mortality (participants affected / at risk) | 3/15 | 0/5
Serious Adverse Events (participants affected / at risk) | 7/15 | 0/5
Other Adverse Events (participants affected / at risk) | 0/15 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HMB-DMR-HA (N=15) | HMB-DM-CEM (N=5)
Surgical infection (Surgical and medical procedures) | 2 (2) | 0 (0)
Intra-prosthetic dislocation (Product Issues) | 1 (1) | 0 (0)
fall and fracture of the operated area (Vancouver class: A) (Surgical and medical procedures) | 1 (1) | 0 (0)
Other (General disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-16): https://cdn.clinicaltrials.gov/large-docs/26/NCT04209426/Prot_SAP_000.pdf